CLINICAL TRIAL: NCT01867723
Title: Improving Symptom Management for Cancer Patients and Their Caregivers Through Internet Support: A Randomized Clinical Trial
Brief Title: Improving Symptom Management for Cancer Patients and Their Caregivers Through Internet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Oslo University Hospital, Center for Shared Decision Making and Collaborative Care Research, Oslo University Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 6.2008.547
Record Dates: First submitted 2012-03-06; First posted 2013-06-04 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Fatigue
Keywords: Cancer internet support program
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet communication application (Experimental): Experiment 1 Effect of internet support program on cancer patients and their caregivers
  Interventions: Other: Internet communication application
- Control group (No Intervention): Control group get usual care

INTERVENTIONS:
Other: Internet communication application — Intervention 1 Effect of internet support program will be tested on cancer patients and their family caregivers No intervention
  Arms: Internet communication application

SUMMARY:
Being diagnosed and treated for cancer is usually associated with severe side effects and symptoms. Cancer patients can have difficulty to manage the symptoms as a result of treatment which may cause i) an interruption or cessation of cancer treatment ii) can have a negative impact on patients' quality of life (QoL). Family caregivers (FCs) of cancer patients are often the primary source of social and emotional support for patients, and play major roles in how well patients manage with the consequences of illness and treatment. Thus, FCs are clinically important, since supporting FCs indirectly supports patients.

To help both cancer patients and their FCs to manage their symptoms, our center has developed WebChoice now called Connect, an internet based support system that extends traditional health services into cancer patients' homes. Connect provides individualized symptom management support, illness relevant information, and communication with a clinical nurse specialist in cancer care, as well as with other cancer patients and their FCs over the Internet. The objectives of this interdisciplinary research project are to test main and interaction effects of providing Connect to patients, to FCs or both simultaneously on 1) primary patient outcomes in terms of symptom distress, QoL, depression, fatigue and sleep 2) Primary FC outcomes in terms of symptom distress, QoL, depression, fatigue, sleep and FC burden 3) Secondary, or intermediate, patient and FC outcomes in terms of self-efficacy social support, and self-reported health care utilization.

DETAILED DESCRIPTION:
Cancer patients often experience multiple symptoms due to the illness itself and its treatment. Failure to detect and relieve patients' symptoms can have deleterious effects on patients [1]. To adequately help patients, it is important to understand how symptoms vary and co-vary during different phases of patients' illness trajectory. A major limitation in previous studies of symptoms in patients undergoing cancer treatment is that they have not evaluated symptom changes over time during and how changes in one or more symptom influence patients QoL. Furthermore, compelling evidence exist that cancer patients do not receive adequate symptom management or palliative care during the course of their illness [2-4].

A barrier to appropriate symptom management is the lack of interventions that support patients effectively in symptom management and self-management. Within the current health system, patients get limited help with their symptoms and health problems. This problem is accentuated by short hospital stays or consultations. Side-effects of treatment usually are at their worst after discharge from the hospital, and patients spend most of the time at home, leaving them with considerable symptom distress without much assistance. To overcome these problems, the Center for Shared Decision Making (CSDM) and Collaborative Care Research at Olso University Hospital (OUS) has developed WebChoice now called Connect, an Internet based support system that extends traditional health services into cancer patients' homes. Connect provides individualized symptom management support, illness relevant information, and communication with a clinical nurse specialist (CNS) in cancer care, as well as with other cancer patients over the Internet. v has been tested in an RCT funded by the Norwegian Cancer Society with breast and prostate cancer patients nationwide. Results from this RCT and other previous studies on Connect components demonstrate significant improvements in patient-centered care [5-7] and patient outcomes in terms of less symptom distress of depression. Also patients with access to WebChoice maintained self-efficacy and health related quality of life over time while the control group deteriorated significantly. (under review). Therefore, an important next step and aim of this study is to expand and test Connect in the following, to benefit a larger group of patients.

Research has repeatedly shown that FCs of cancer patients experience many problems, symptoms and burden [8]. However, the relationship between patient and FCs symptoms and problems is not yet sufficiently understood. Affecting one may also affect the other, and interventions that support FCs could also support patients and vice versa, reducing symptom distress [9]. Therefore, we will extend Connect to support cancer patients and their FCs, and test its effects on patient and FC outcomes.

Thus the specific aims for Phase II of this project are to:

1. Develop and test the effects of an extended Connect module to support (1) cancer patients and (2) their FCs on patient and FC outcomes.

Research Questions:

Following cancer patients and their FCs with 3 repeated measures over 6 months, this study will test main and interaction effects of providing Connect to patients, to FCs or both simultaneously on:

* Primary patient outcomes in terms of symptom distress, HRQoL, depression, fatigue and sleep.
* Primary FC outcomes in terms of symptom distress, QoL, depression, fatigue, sleep and care giver burden.
* Secondary, or intermediate, patient and FC outcomes in terms of self-efficacy, social support, and self-reported health care utilization.
* To better understand how these effects may occur, we will explore relationships between primary patient and FC outcomes; and how primary and secondary outcomes vary and co-vary across experimental conditions. Additional research questions are:
* How do patients and FCs use Connect? What is the frequency of use and which components are most used?
* What are patients' and FCs perceptions of usefulness and ease of use of Connect?

ELIGIBILITY:
Inclusion Criteria:

* diagnosed and treated for cancer;
* > 18 years of age,
* able to read/write/speak Norwegian,
* written informed consent, and
* have a FC who is willing to participate. FCs will be the individual the patient identifies as being most involved in their care.

Exclusion Criteria:

* Patients received cranial radiation or who have brain metastasis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Actual)
Dates: Start 2012-04; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change from the Baseline in severity and duration of HRQoL | Baseline, 3 og 6 months
Change from the baseline in severity and duration of depression | Baseline, 3 and 6 months
Change from the Baseline in severity and duration of fatigue | Baseline, 3 and 6 months
Change from the baseline in severity and duration of sleep disorder | Baseline, 3 and 6 months

SECONDARY OUTCOMES:
Change from baseline in self-efficacy | Baseline and at 3 and 6 months
Change from baseline in social support | Baseline, 3 and 6 months
Change from baseline in self-reported health care utilization | Baseline, 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Ruland, PHD, Principal Investigator — Oslo University Hospital- Raikshospitalet
Locations (1):
- Oslo University Hospital, Oslo, Oslo County, Norway

REFERENCES:
- [Background] Sygna K, Johansen S, Ruland CM. Recruitment challenges in clinical research including cancer patients and their caregivers. A randomized controlled trial study and lessons learned. Trials. 2015 Sep 25;16:428. doi: 10.1186/s13063-015-0948-y. Erratum In: Trials. 2016 Mar 10;17(1):133. doi: 10.1186/s13063-016-1276-6. PMID 26407547